CLINICAL TRIAL: NCT04199104
Title: A Phase 3, Randomized, Placebo-controlled, Double-blind Clinical Study of Pembrolizumab (MK-3475) With or Without Lenvatinib (E7080/MK-7902) to Evaluate the Safety and Efficacy of Pembrolizumab and Lenvatinib as 1L Intervention in a PD-L1 Selected Population of Participants With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (R/M HNSCC) (LEAP-010).
Brief Title: A Study of Pembrolizumab (MK-3475) With or Without Lenvatinib (E7080/MK-7902) as First Line (1L) Intervention in a Programmed Cell Death-ligand 1 (PD-L1) Selected Population With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (R/M HNSCC) (MK-7902-010) (KEYNOTE-010)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7902-010; MK-7902-010 (Other: MSD); LEAP-10 (Other: MSD); 205240 (Registry Identifier: JAPIC-CTI); 2019-003717-34 (EudraCT Number)
Record Dates: First submitted 2019-12-12; First posted 2019-12-13 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: head and neck squamous cell carcinoma; pembrolizumab; lenvatinib; PD-L1
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — lenvatinib; pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab with Lenvatinib (Experimental): Participants receive lenvatinib 20 mg orally once a day (QD) plus pembrolizumab 200 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W). Pembrolizumab will be administered for up to 35 cycles (approximately 24 months). Lenvatinib will be administered until progressive disease or unacceptable toxicity.
  Interventions: Drug: Lenvatinib; Biological: Pembrolizumab
- Pembrolizumab with Placebo (Active Comparator): Participants receive lenvatinib-matching placebo orally once a day (QD) plus pembrolizumab 200 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W). Pembrolizumab will be administered for up to 35 cycles (approximately 24 months).
  Interventions: Biological: Pembrolizumab; Drug: Placebo

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib, 20 mg (two 10-mg oral capsules) administered QD
  Other Names: E7080; MK-7902; LENVIMA®
  Arms: Pembrolizumab with Lenvatinib
Biological: Pembrolizumab — Pembrolizumab (MK-3475), 200 mg, every 3 weeks (Q3W) by intravenous (IV) infusion for up to 35 3-week cycles
  Other Names: MK-3475; Keytruda®
Drug: Placebo — Lenvatinib-matching placebo, oral capsules, administered once daily (QD)
  Arms: Pembrolizumab with Placebo

SUMMARY:
This is a study of pembrolizumab (MK-3475) with or without lenvatinib (E7080/MK-7902) as a first line intervention in a PD-L1 selected population with participants with recurrent or metastatic head and neck squamous cell carcinoma.

Hypotheses include:

* Pembrolizumab + lenvatinib is superior to pembrolizumab + placebo with respect to Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by blinded independent central review (BICR).
* Pembrolizumab + lenvatinib is superior to pembrolizumab + placebo with respect to Progression Free Survival (PFS) per RECIST 1.1 as assessed by BICR.
* Pembrolizumab + lenvatinib is superior to pembrolizumab + placebo with respect to overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Has histologically confirmed diagnosis of R/M HNSCC that is considered incurable by local therapies.

Note: Participants with newly-diagnosed HNSCC must be M1/Stage IV.

* Has a primary tumor location of oropharynx, oral cavity, hypopharynx, or larynx.

Note: Primary tumor site of nasopharynx (any histology) or unknown primary tumor (including p16+ unknown primary) are not eligible.

Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. If the contraception requirements in the local label for any of the study interventions is more stringent than the requirements above, the local label requirements are to be followed.

* Male participants agree to use approved contraception during the treatment period for at least 7 days after the last dose of lenvatinib/placebo, or refrain from heterosexual intercourse during this period
* Female participants are not pregnant or breastfeeding, and are not a woman of childbearing potential (WOCBP), OR are a WOCBP that agrees to use contraception during the treatment period (or 14 days prior to the initiation of study treatment for oral contraception) and for at least 120 days post pembrolizumab, or 30 days post lenvatinib/placebo, whichever occurs last
* Has measurable disease per RECIST 1.1 as assessed by BICR. Note: Lesions situated in a previously irradiated area are considered measurable if progression has been shown in such lesions.
* Participants with oropharyngeal cancer must have results from testing of human papillomavirus HPV status.
* Has an Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 1.
* Have adequately controlled blood pressure with or without antihypertensive medications.
* Has adequate organ function.

Exclusion Criteria:

* Has a history of any contraindication or has a severe hypersensitivity to any components of pembrolizumab (≥Grade 3) or lenvatinib.
* Has pre-existing ≥Grade 3 gastrointestinal or non-gastrointestinal fistula.
* Has a history of a gastrointestinal condition or procedure that, in the opinion of the investigator, may affect oral study drug absorption.
* Has clinically significant cardiovascular impairment within 12 months of the first dose of study intervention, such as history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or cerebrovascular accident/transient ischemic attack (TIA)/stroke, cardiac revascularization, or cardiac arrhythmia associated with hemodynamic instability.
* Has disease that is suitable for local therapy administered with curative intent.
* Had PD within 6 months of completion of curatively intended systemic treatment for locoregionally advanced HNSCC.
* Has had major surgery within 3 weeks before to first dose of study interventions.
* Has difficulty swallowing capsules or ingesting a suspension orally or by a feeding tube.
* Has received prior therapy with lenvatinib or pembrolizumab.
* Received last dose of systemic therapy for locoregionally advanced disease less than 6 months before signing consent.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137).
* Has received prior systemic anticancer therapy including investigational agents within 4 weeks before randomization.
* Has received prior radiotherapy within 2 weeks of start of study intervention.
* Has received a live vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
* Received an investigational agent or has used an investigational device within 4 weeks prior to study intervention-administration.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study intervention.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.

Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.

* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has an active autoimmune disease that has required systemic treatment in past 2 years. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid) is allowed.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy. (e.g., tuberculosis, known viral or bacterial infections, etc.).
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has a known history of hepatitis B (defined as HBsAg reactive) or known active hepatitis C virus (defined as HCV ribonucleic acid (RNA) [qualitative] is detected) infection.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study intervention.
* Has had an allogenic tissue/solid organ transplant.
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (152):
- United States (26):
  - California Cancer Associates for Research & Excellence ( Site 0025), Fresno, California
  - California Cancer Associates for Research & Excellence ( Site 0059), San Marcos, California
  - University of Colorado Cancer Center ( Site 0023), Aurora, Colorado
  - University of Connecticut Health Center ( Site 0020), Farmington, Connecticut
  - Memorial Regional Hospital-Memorial Cancer Institute ( Site 0069), Hollywood, Florida
  - Georgia Cancer Center at Augusta University ( Site 0013), Augusta, Georgia
  - Northwest Georgia Oncology Centers PC ( Site 0028), Marietta, Georgia
  - University of Kansas Cancer Center ( Site 0033), Westwood, Kansas
  - University of Louisville, James Graham Brown Cancer Center ( Site 0045), Louisville, Kentucky
  - Dana Farber Cancer Institute ( Site 0019), Boston, Massachusetts
  - University of Michigan ( Site 0064), Ann Arbor, Michigan
  - Karmanos Cancer Institute ( Site 0054), Detroit, Michigan
  - Henry Ford Health System ( Site 0001), Detroit, Michigan
  - Washington University School of Medicine ( Site 0060), St Louis, Missouri
  - St. Vincent Frontier Cancer Center ( Site 0008), Billings, Montana
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists ( Site 0053), Omaha, Nebraska
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 0002), Hackensack, New Jersey
  - Weill Cornell Medicine New York Presbyterian Hospital ( Site 0040), New York, New York
  - SUNY Upstate Medical University ( Site 0051), Syracuse, New York
  - University of North Carolina- Chapel Hill ( Site 0056), Chapel Hill, North Carolina
  - Duke Cancer Center ( Site 0044), Durham, North Carolina
  - Providence Portland Medical Center ( Site 0048), Portland, Oregon
  - Blue Ridge Cancer Care ( Site 0015), Blacksburg, Virginia
  - Inova Schar Cancer Institute ( Site 0009), Fairfax, Virginia
  - Cancer Care Northwest ( Site 0017), Spokane Valley, Washington
  - University of Wisconsin- Madison Carbone Cancer Center ( Site 0006), Madison, Wisconsin
- Australia (3):
  - Chris OBrien Lifehouse ( Site 1002), Camperdown, New South Wales
  - St George Hospital ( Site 1001), Kogarah, New South Wales
  - Royal Adelaide Hospital ( Site 1004), Adelaide, South Australia
- Brazil (7):
  - Oncocentro Ceara ( Site 0412), Fortaleza, Ceará
  - Fundacao Sao Francisco Xavier ( Site 0409), Ipatinga, Minas Gerais
  - ELO Pesquisa Clinica ( Site 0405), Maringá, Paraná
  - Hospital de Passo Fundo ( Site 0401), Passo Fundo, Rio Grande do Sul
  - Clinica LACKS ( Site 0402), Pelotas, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceição-Centro Integrado de Pesquisa em Oncologia ( Site 0414), Porto Alegre, Rio Grande do Sul
  - A.C. Camargo Cancer Center ( Site 0407), São Paulo
- Canada (3):
  - Princess Margaret Cancer Centre ( Site 0200), Toronto, Ontario
  - McGill University Health Centre ( Site 0206), Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus ( Site 0, Québec, Quebec
- China (20):
  - Beijing Cancer Hospital ( Site 3314), Beining, Beijing Municipality
  - Peking Union Medical College Hospital ( Site 3304), Bejiing, Beijing Municipality
  - Chongqing Cancer Hospital ( Site 3327), Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital ( Site 3326), Fuzhou, Fujian
  - Guangxi Medical University Affiliated Tumor Hospital ( Site 3322), Nanning, Guangxi
  - Guizhou Cancer Hospital ( Site 3330), Guiyang, Guizhou
  - The Third Affiliated Hospital of Harbin Medical University ( Site 3302), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 3309), Zhengzhou, Henan
  - Wuhan Union hospital Cancer Center ( Site 3307), Wuhan, Hubei
  - Tongji Hospital Tongji Medical,Science & Technology ( Site 3316), Wuhan, Hubei
  - Hunan Cancer Hospital ( Site 3311), Changsha, Hunan
  - Xiangya Hospital of Central South University ( Site 3305), Changsha, Hunan
  - Jiangxi Cancer Hospital ( Site 3313), Nanchang, Jiangxi
  - Jilin Cancer Hospital ( Site 3310), Changchun, Jilin
  - The First Affiliated Hospital of Xi an Jiaotong University ( Site 3328), Xi'an, Shaanxi
  - Fudan University Shanghai Cancer Center ( Site 3324), Shanghai, Shanghai Municipality
  - Shanghai East Hospital ( Site 3300), Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University ( Site 3308), Chengdu, Sichuan
  - Tianjin Medical University Cancer Hospital ( Site 3312), Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital ( Site 3303), Hangzhou, Zhejiang
- France (5):
  - Centre Leon Berard ( Site 1901), Lyon, Auvergne
  - Hopital de la Timone ( Site 1903), Marseille, Bouches-du-Rhone
  - Hopital Foch ( Site 1905), Suresnes, Hauts-de-Seine
  - Centre Henri Becquerel ( Site 1904), Rouen, Seine-Maritime
  - Gustave Roussy ( Site 1906), Villejuif, Val-de-Marne
- Germany (8):
  - Universitaetsklinikum Tuebingen ( Site 2108), Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Ulm ( Site 2102), Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Regensburg ( Site 2100), Regensburg, Bavaria
  - Universitaetsklinikum Frankfurt ( Site 2107), Frankfurt am Main, Hesse
  - KRH Klinikum Siloah ( Site 2103), Hanover, Lower Saxony
  - Universitaetsklinikum Koeln ( Site 2111), Cologne, North Rhine-Westphalia
  - Universitätsklinikum Leipzig-Department for ENT ( Site 2106), Leipzig, Saxony
  - Charite Universitätsmedizin Berlin Campus Benjamin Franklin ( Site 2112), Berlin
- Hungary (6):
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Egyetemi Okta-Klinikai Onkológiai és Sugárterápiás Ce, Miskolc, Borsod-Abauj Zemplen county
  - Szegedi Egyetem Szent-Gyorgyi Albert Klinikai Kozpont ( Site 2207), Szeged, Csongrád megye
  - Jasz Nagykun Szolnok Megyei Hetenyi Geza Korhaz Rendelointezet ( Site 2200), Szolnok, Jász-Nagykun-Szolnok
  - Uzsoki Utcai Korhaz ( Site 2201), Budapest, Vas County
  - Orszagos Onkologiai Intezet ( Site 2202), Budapest
  - Debreceni Egyetem Klinikai Kozpont ( Site 2206), Debrecen
- Italy (6):
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia ( Site 2402), Brescia
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 2400), Milan
  - IEO Istituto Europeo di Oncologia ( Site 2406), Milan
  - ASST Santi Paolo e Carlo - Presidio Ospedaliero San Paolo ( Site 2405), Milan
  - Istituto Oncologico Veneto ( Site 2404), Padua
  - ASL Liguria 2 - Ospedale San Paolo ( Site 2401), Savona
- Japan (14):
  - Aichi Cancer Center Hospital ( Site 1113), Nagoya, Aichi-ken
  - Nagoya University Hospital ( Site 1106), Nagoya, Aichi-ken
  - Chiba cancer center ( Site 1110), Chiba, Chiba
  - National Cancer Center Hospital East ( Site 1100), Kashiwa, Chiba
  - Hyogo Cancer Center ( Site 1112), Akashi, Hyōgo
  - Kagawa University Hospital ( Site 1108), Kita-gun, Kagawa-ken
  - Yokohama City University Hospital ( Site 1104), Yokohama, Kanagawa
  - Kindai University Hospital ( Site 1107), Sayama, Osaka
  - Shizuoka Cancer Center Hospital and Research Institute ( Site 1105), Sunto-gun, Shizuoka
  - National Hospital Organization Kyushu Medical Center ( Site 1111), Fukuoka
  - Hiroshima University Hospital ( Site 1109), Hiroshima
  - National Cancer Center Hospital ( Site 1102), Tokyo
  - The Cancer Institute Hospital of JFCR ( Site 1103), Tokyo
  - Tokyo Medical and Dental University Hospital ( Site 1101), Tokyo
- Mexico (5):
  - Cryptex Investigación Clínica S.A. de C.V. ( Site 0608), Cuauhtémoc, Mexico City, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez" ( Site 0602), Monterrey, Nuevo León
  - Christus Muguerza Clinica Vidriera ( Site 0607), Monterrey, Nuevo León
  - Centro de Investigacion y Avances Medicos Especializados -CIAME ( Site 0604), Cancún, Quintana Roo
  - Oaxaca Site Management Organization S.C. ( Site 0603), Oaxaca City
- Peru (5):
  - Instituto Nacional de Enfermedades Neoplasicas ( Site 0701), Lima, Muni Metro de Lima
  - Hospital Nacional Guillermo Almenara Irigoyen ( Site 0700), Lima
  - Hospital Nacional Edgardo Rebagliati Martins ( Site 0702), Lima
  - Hospital Nacional Arzobispo Loayza ( Site 0703), Lima
  - Hospital Nacional Cayetano Heredia ( Site 0704), Lima
- Poland (8):
  - Przychodnia Lekarska Komed ( Site 2500), Konin, Greater Poland Voivodeship
  - Szpital Kliniczny im. Heliodora Swiecickiego Uniwers Medyczn ( Site 2509), Poznan, Greater Poland Voivodeship
  - Centrum Onkologii im prof Franciszka Lukaszczyka ( Site 2508), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie ( Site 2502), Krakow, Lesser Poland Voivodeship
  - Dolnoslaskie Centrum Onkologii. ( Site 2507), Wroclaw, Lower Silesian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworow Glowy i Szyi ( Site, Warsaw, Masovian Voivodeship
  - Szpital Morski im. PCK. Szpitale Pomorskie Sp. Z o.o ( Site 2504), Gdynia, Pomeranian Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach ( Site 2506), Gliwice, Silesian Voivodeship
- Russia (4):
  - Altay Regional Oncology Dispensary ( Site 2611), Barnaul, Altayskiy Kray
  - FSCC FMBA of Russia ( Site 2603), Moscow, Moscow
  - Republican Clinical Oncology Dispensary of Tatarstan MoH ( Site 2609), Kazan', Tatarstan, Respublika
  - Yaroslavl Regional SBIH Clinical Oncology Hospital ( Site 2605), Yaroslavl, Yaroslavl Oblast
- South Korea (6):
  - Chonnam National University Hwasun Hospital ( Site 1202), Hwasun-gun, Jeonranamdo
  - Seoul National University Bundang Hospital ( Site 1205), Seongnam-si, Kyonggi-do
  - Ajou University Hospital ( Site 1200), Suwon, Kyonggi-do
  - Asan Medical Center ( Site 1201), Songpa-gu, Seoul
  - Keimyung University Dongsan Hospital ( Site 1203), Daegu, Taegu-Kwangyokshi
  - The Catholic University of Korea Eunpyeong St Mary s Hospital ( Site 1204), Seoul
- Spain (6):
  - Hospital Duran i Reynals ( Site 2701), L'Hospitalet de Llobregat, Barcelona
  - H.U. Vall de Hebron ( Site 2700), Barcelona
  - Hospital Universitario 12 de Octubre ( Site 2702), Madrid
  - Hospital Universitario La Paz ( Site 2706), Madrid
  - Hospital de Valme ( Site 2705), Seville
  - Hospital Clinico Universitario Lozano Blesa ( Site 2703), Zaragoza
- Taiwan (5):
  - National Cheng Kung University Hospital ( Site 1603), Dawan, Tainan
  - Chang Gung Medical Foundation. Kaohsiung Branch ( Site 1604), Kaohsiung City
  - National Taiwan University Hospital ( Site 1600), Taipei
  - MacKay Memorial Hospital ( Site 1602), Taipei
  - Taipei Veterans General Hospital ( Site 1601), Taipei
- Turkey (Türkiye) (7):
  - Hacettepe Universitesi Tip Fakultesi ( Site 2805), Ankara
  - Ankara Sehir Hastanesi ( Site 2802), Ankara
  - Trakya Universitesi Tip Fakultesi ( Site 2801), Edirne
  - Medipol Universite Hastanesi ( Site 2800), Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi ( Site 2804), Izmir
  - Medical Park Izmir Hospital ( Site 2807), Izmir
  - Inonu Universitesi Turgut Ozal Tip Merkezi ( Site 2803), Malatya
- United Kingdom (8):
  - Aberdeen Royal Infirmary ( Site 2905), Aberdeen, Aberdeen City
  - Guy's Hospital in London ( Site 2908), London, London, City of
  - Royal Marsden NHS Foundation Trust ( Site 2910), London, London, City of
  - Mount Vernon Cancer Centre ( Site 2902), Northwood, London, City of
  - Royal Marsden Hospital ( Site 2904), Sutton, London, City of
  - Nottingham City Hospital ( Site 2907), Nottingham, Nottinghamshire
  - Taunton and Somerset Hospital ( Site 2900), Taunton, Somerset
  - Christie NHS Foundation Trust ( Site 2903), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Taylor MH, Schmidt EV, Dutcus C, Pinheiro EM, Funahashi Y, Lubiniecki G, Rasco D. The LEAP program: lenvatinib plus pembrolizumab for the treatment of advanced solid tumors. Future Oncol. 2021 Feb;17(6):637-648. doi: 10.2217/fon-2020-0937. Epub 2020 Dec 10. PMID 33300372
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab + Lenvatinib: Participants were administered Pembrolizumab 200mg by intravenous IV infusion on Day 1 of each 21-day cycle (Q3W) plus Lenvatinib 20 mg orally once a day (QD)
- Pembrolizumab + Placebo: Participants were administered lenvatinib-matching placebo orally once a day (QD) plus pembrolizumab 200 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W).
Period: Overall Study
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Started | 256 | 255
Treated | 254 | 253
Received Second Course | 2 | 0
Completed | 0 | 0
Not Completed | 256 | 255
Not completed — Death | 148 | 134
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Participants Ongoing | 103 | 116

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo | Total
Number analyzed (Participants) | 256 | 255 | 511
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.0 (8.8) | 62.7 (9.6) | 63.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 42 | 79
  Male | 219 | 213 | 432
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 43 | 76
  Not Hispanic or Latino | 205 | 198 | 403
  Unknown or Not Reported | 18 | 14 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 7 | 9
  Asian | 67 | 80 | 147
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 168 | 147 | 315
  More than one race | 17 | 19 | 36
  Unknown or Not Reported | 0 | 0 | 0
Programmed Cell Death Ligand 1 (PD-L1) Tumor Expression [Count of Participants; unit: Participants] — Participants were assessed for their PD- L1 tumor expression level by immunohistochemistry assay using tumor tissue from a newly obtained biopsy. PD-L1 expression analyses were restricted to only tumor cells with TPS (tumor proportion scoring) <50% vs ≥50%.
  Participants
    <50% | 192 | 191 | 383
    >=50% | 64 | 64 | 128
Human Papilloma Virus (HPV) Status [Count of Participants; unit: Participants] — HPV status for oropharynx cancer as determined by immunohistochemistry (positive or negative); HPV status for participants without oropharynx cancer (eg, cancers of the oral cavity, hypopharynx and larynx) is considered HPV negative.
  Participants
    Positive | 57 | 58 | 115
    Negative | 199 | 197 | 396
Eastern Cooperative Oncology Group (ECOG Status of 0 vs 1) [Count of Participants; unit: Participants] — Participants were stratified on basis of their ECOG status of 0 vs 1. The ECOG status 0 meant fully active, able to carry on all pre-disease performance without restriction, whereas an ECOG status 1 meant restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature.
  Participants
    ECOG 0 | 122 | 115 | 237
    ECOG 1 | 134 | 140 | 274

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: ORR is defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. The percentage of participants who experienced a CR or PR based on modified RECIST 1.1 is presented.
Time Frame: Up to ~ 37 months
Population: All randomized participants were included from the intention to treat (ITT) participants. Participants were included in the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 256 | 255
Percentage of participants | 46.9 [40.6 to 53.2] | 27.5 [22.1 to 33.4]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Superiority; p = 0.0000019, Miettinen and Nurminen method; point estimate = 19.3, 95% CI 2-sided [11.2 to 27.3]

2. Primary Outcome: Progression Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR).
Description: PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions is also considered PD.
Time Frame: Up to ~ 37 months
Population: All randomized participants included in the ITT participants. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 256 | 255
Months | 7.0 [5.6 to 8.0] | 2.8 [2.6 to 4.1]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Superiority; p = 0.0001129, Regression, Cox; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.55 to 0.83]

3. Primary Outcome: Overall Survival (OS)
Description: OS is the time from randomization to death due to any cause.
Time Frame: Up to ~ 37 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 256 | 255
Months | 15.0 [13.2 to 17.0] | 17.9 [13.8 to 21.6]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Superiority; p = 0.8819584, Regression, Cox; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.91 to 1.45]

4. Secondary Outcome: Duration of Response (DOR)
Description: For participants who demonstrate a confirmed complete response (CR: Disappearance of all target lesions) or confirmed Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until disease progression or death.
Time Frame: Up to ~ 37 months
Population: All randomized participants included in the ITT participants who demonstrated at least a partial response. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 120 | 70
Months | 10.1 [8.3 to 13.9] | NA [11.9 to NA] — Median and upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse.

5. Secondary Outcome: Percentage of Participants Who Experienced an Adverse Event (AE)
Description: An adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to ~ 37 months
Population: Safety analyses was conducted in the all-participants-as-treated (APaT) population, which consisted of all randomized participants who received at least one dose of study treatment. Participants were included in the treatment group corresponding to the study treatment they actually received.
Measure: Number; unit: Percentage of Participants
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 254 | 253
Percentage of Participants | 99.21 | 96.84

6. Secondary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an AE
Description: as for outcome 5
Time Frame: Up to ~ 34 months
Population: Safety analyses was conducted in the APaT population, which consisted of all randomized participants who received at least one dose of study treatment. Participants were included in the treatment group corresponding to the study treatment they actually received.
Measure: Number; unit: Percentage of Participants
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 254 | 253
Percentage of Participants | 43.7 | 15.02

ADVERSE EVENTS:
Time Frame: Up to ~ 37 months
Description: All-cause mortality (ACM) was analyzed in all randomized participants. Safety analyses were conducted in all randomized participants who received at least 1 dose of study intervention. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Thus, MedDRA 26.0 preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to the drug are excluded.
Groups:
- Pembrolizumab + Lenvatinib First Course: Participants were administered Pembrolizumab 200mg by intravenous IV infusion on Day 1 of each 21-day cycle (Q3W) plus Lenvatinib 20 mg orally once a day (QD).
- Pembrolizumab + Lenvatinib Second Course: Pembrolizumab was administered 200mg by intravenous IV infusion on Day 1 of each 21-day cycle (Q3W) for 17 cycles (~ 1 year) and Lenvatinib/Placebo at the last dose level was continued during second course at investigators discretion.
Arm/Group | Pembrolizumab + Lenvatinib First Course | Pembrolizumab + Placebo | Pembrolizumab + Lenvatinib Second Course
All-Cause Mortality (participants affected / at risk) | 152/256 | 138/255 | 0/2
Serious Adverse Events (participants affected / at risk) | 152/254 | 89/253 | 0/2
Other Adverse Events (participants affected / at risk) | 244/254 | 221/253 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Lenvatinib First Course (N=254) | Pembrolizumab + Placebo (N=253) | Pembrolizumab + Lenvatinib Second Course (N=2)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 (0) | 1 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 2 (2) | 0 (0)
Hypercalcaemia of malignancy (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 7 (8) | 6 (6) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Salivary duct inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 6 (6) | 3 (3) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 2 (2) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 3 (3) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fournier's gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Necrotising soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Perineal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 20 (24) | 12 (13) | 0 (0)
Pneumonia acinetobacter (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 7 (8) | 4 (4) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia necrotising (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Stoma site infection (Infections and infestations) | 2 (5) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Radiation necrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (6) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Fulminant type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (3) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Oral haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (14) | 8 (9) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Autonomic dysreflexia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Diabetic hyperosmolar coma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 3 (3) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Autoimmune lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Lenvatinib First Course (N=254) | Pembrolizumab + Placebo (N=253) | Pembrolizumab + Lenvatinib Second Course (N=2)
Anaemia (Blood and lymphatic system disorders) | 65 (95) | 51 (73) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 6 (6) | 2 (2) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 19 (22) | 10 (10) | 0 (0)
Hypothyroidism (Endocrine disorders) | 124 (145) | 43 (49) | 0 (0)
Bowel movement irregularity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 56 (73) | 46 (55) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 71 (111) | 33 (45) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 17 (18) | 18 (19) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 14 (22) | 3 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 35 (39) | 14 (15) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 62 (83) | 25 (27) | 0 (0)
Oral pain (Gastrointestinal disorders) | 29 (34) | 6 (7) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 53 (73) | 12 (12) | 0 (0)
Vomiting (Gastrointestinal disorders) | 33 (48) | 14 (16) | 0 (0)
Asthenia (General disorders) | 26 (32) | 25 (30) | 1 (1)
Fatigue (General disorders) | 80 (91) | 41 (44) | 1 (1)
Mucosal inflammation (General disorders) | 25 (35) | 7 (10) | 0 (0)
Pyrexia (General disorders) | 20 (22) | 19 (24) | 0 (0)
COVID-19 (Infections and infestations) | 16 (17) | 13 (13) | 0 (0)
Pneumonia (Infections and infestations) | 25 (26) | 11 (12) | 0 (0)
Urinary tract infection (Infections and infestations) | 13 (16) | 13 (15) | 0 (0)
Alanine aminotransferase increased (Investigations) | 36 (49) | 21 (27) | 0 (0)
Amylase increased (Investigations) | 14 (20) | 14 (21) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 37 (56) | 23 (30) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 13 (15) | 19 (21) | 0 (0)
Blood bilirubin increased (Investigations) | 17 (20) | 7 (9) | 0 (0)
Blood creatinine increased (Investigations) | 26 (27) | 5 (6) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 16 (21) | 7 (7) | 0 (0)
Lipase increased (Investigations) | 30 (36) | 17 (28) | 0 (0)
Lymphocyte count decreased (Investigations) | 30 (57) | 20 (33) | 0 (0)
Platelet count decreased (Investigations) | 31 (42) | 8 (13) | 0 (0)
Weight decreased (Investigations) | 65 (72) | 39 (41) | 0 (0)
White blood cell count decreased (Investigations) | 16 (33) | 10 (16) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 57 (69) | 23 (24) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 11 (13) | 18 (20) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 (22) | 11 (12) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 18 (20) | 7 (8) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 34 (45) | 23 (25) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 22 (29) | 9 (11) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 22 (29) | 7 (9) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 44 (71) | 28 (36) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 14 (16) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 40 (52) | 18 (25) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (5) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 18 (18) | 8 (9) | 0 (0)
Dizziness (Nervous system disorders) | 13 (18) | 8 (8) | 0 (0)
Headache (Nervous system disorders) | 32 (37) | 16 (16) | 0 (0)
Insomnia (Psychiatric disorders) | 25 (27) | 12 (13) | 0 (0)
Haematuria (Renal and urinary disorders) | 13 (18) | 7 (11) | 0 (0)
Proteinuria (Renal and urinary disorders) | 62 (112) | 16 (17) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 40 (44) | 23 (25) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 23 (26) | 4 (4) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 (31) | 14 (14) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 10 (18) | 10 (12) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 28 (32) | 8 (8) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 10 (10) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 6 (6) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 15 (15) | 8 (8) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 36 (51) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 27 (32) | 29 (42) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 34 (46) | 23 (26) | 0 (0)
Hypertension (Vascular disorders) | 117 (204) | 24 (36) | 0 (0)
Hypotension (Vascular disorders) | 14 (15) | 7 (8) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/04/NCT04199104/Prot_SAP_000.pdf